CLINICAL TRIAL: NCT05074082
Title: PelvEx 8: Perineal Flap Reconstruction Following Surgery for Advanced Pelvic Malignancy
Brief Title: Perineal Flap Reconstruction Following Surgery for Advanced Pelvic Malignancy
Status: Completed | Type: Observational
Sponsor: St Vincent's University Hospital, Ireland (Other)
Collaborators: PelvEx (Unknown)
Responsible Party: Principal Investigator, Professor Des Winter, Professor Desmond C Winter, St Vincent's University Hospital, Ireland
Other Study IDs: PelvEx 8
Record Dates: First submitted 2021-09-29; First posted 2021-10-12 (Actual); Last update posted 2023-03-31 (Actual); Status verified 2023-03

CONDITIONS: Pelvic Cancer; Rectal Cancer; Flap Disorder; Flap Ischemia; Flap Necrosis; Perioperative Complication
MeSH Terms: conditions — Pelvic Neoplasms; Rectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Flap reconstruction: Patients who had a flap formation as part of a multi-visceral extended resection for advanced pelvic (rectal, urological, gynaecological, sarcomatous origin) malignancy
  Interventions: Procedure: Flap reconstruction

INTERVENTIONS:
Procedure: Flap reconstruction — Formation of a (myo-/fascio-)cutaneous flap for repair of a skin and soft tissue defect
  Other Names: VRAM flap; ORAM flap; Gracilis flap; IGAP flap; Omental flap

SUMMARY:
Flap reconstruction is utilised increasingly for repair of skin and soft tissue defects following pelvic exenteration. Many methods have been proposed but the outcomes associated with each remain largely unknown and the choice dependant on surgeon preference and patient/ disease characteristics. This review sought to assess the preferred methods for perineal reconstruction following pelvic exenteration by retrospectively assessing the outcomes associated with each at an international, multi-centre level.

DETAILED DESCRIPTION:
Locally advanced pelvic malignancies pose numerous technical difficulties to oncological surgeons, particularly where extended resections are performed. The repair of skin and soft tissue defects after radical resections are among the most challenging. Complications related to wound healing are among the most commonly encountered. They can increase rates of infection in the short-term and often become chronic and difficult to treat. This is particularly relevant in the context of pelvic exenteration, where a larger dead space confers a greater risk of deep perineal wound infection and prior (chemo)radiotherapy impairs tissue quality with suboptimal healing. Primary closure may also lead to higher tension closure where there is a bigger defect, further compounding risk. The first meta-analysis comparing primary closure to flap closure noted a two-fold increased risk of overall wound complications with primary closure (1).

With increasingly extensive procedures being carried out in dedicated centres over recent decades, the use of flap reconstruction for closure of pelvic oncological defects has increased significantly. Perineal reconstruction has been shown to decrease the incidence the wound of break-down as well as the need for a secondary repair of dehiscence (2). More importantly, these complications have been shown to be decreasing over time, suggesting improved techniques and/or better perioperative care. However, this is countered by an increase in the incidence of overall minor complications and the possibility of flap failure necessitating a return to theatre. Flap formation is a morbid procedure in its own right and can involve more intensive nursing care and restrict a patient's mobility after pelvic exenteration, further predisposing to post-operative complications and increasing length-of-stay.

The Vertical Rectus Abdominis Muscle (VRAM) flap remains one of the most commonly used and is considered by some to be the gold standard. However, a wide variety of methods have been proposed but exactly how often each is employed and with what outcomes remains largely unknown and is of great interest to surgeons involved in pelvic reconstruction. This review sought to assess the preferred methods for perineal reconstruction following pelvic exenteration by retrospectively assessing the outcomes associated with each at an international, multi-centre level.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven locally advanced or recurrent pelvic cancer (all subtypes - Rectal, Urological, Gynaecological, Sarcoma)
* Aged over 18 years
* Undergoing a multi-visceral extended pelvic resection and requiring reconstruction of a skin and soft tissue defect as a result
* Time period: 1st July 2016 - 1st July 2021

Exclusion Criteria:

* Strong evidence of metastatic or peritoneal disease
* No immediate flap reconstruction performed at time of extended pelvic resection/pelvic exenteration, or flap reconstruction performed as a delayed procedure or as a response to a complication of prior pelvic exenteration
* Insufficient patient follow-up (Minimum of 30 days)

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients undergoing flap reconstruction of a skin or soft tissue defect as part of a multi-visceral extended resection for pelvic malignancy.
Sampling Method: Non-Probability Sample
Enrollment: 883 (Actual)
Dates: Start 2021-07-31 (Actual); Primary Completion 2022-07-01 (Actual); Study Completion 2023-03-01 (Actual)

PRIMARY OUTCOMES:
Flap reconstruction by procedure | July 2016 - July 2021
  Type of flap formation
Morbidity | July 2016 - July 2021
  Short-term (<30 days) outcomes associated with each type
Clavien-Dindo grade III or greater | July 2016 - July 2021
  Need for re-intervention by flap type
Major flap dehiscence | July 2016 - July 2021
  By flap type

SECONDARY OUTCOMES:
Length of stay | July 2016 - July 2021
  Duration of post-operative hospital stay by flap type

CONTACTS AND LOCATIONS:
Overall Officials: Desmond C Winter, MD, Principal Investigator — St. Vincent's Healthcare Group
Locations (1):
- St. Vincent's Hospital, Dublin, Ireland

IPD SHARING:
Plan to Share IPD: No